CLINICAL TRIAL: NCT00218439
Title: Smoking, Antidepressants, and Response to Mental Stress
Brief Title: Effect of Paroxetine on Smokers' Cardiovascular Response to Stress - 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0310M52790; K23DA017307-01 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Tobacco Use Disorder
Keywords: Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Active medication for 4 weeks followed by placebo for 4 weeks
  Interventions: Drug: Paroxetine; Drug: Placebo
- 2 (Experimental): Placebo for 4 weeks followed by active for 4 weeks
  Interventions: Drug: Paroxetine; Drug: Placebo

INTERVENTIONS:
Drug: Paroxetine — 10 mg for 1 week followed by 20 mg for 3 weeks
Drug: Placebo

SUMMARY:
Smokers report that they often smoke cigarettes during stressful times. The combined effect of smoking and exposure to stress leads to exaggerated increases in blood pressure, heart rate and other measures of stress response. This combination may result in greater cardiovascular harm than either smoking or stress alone. The purpose of this study is to determine the effects of paroxetine on the response to stress after smoking.

DETAILED DESCRIPTION:
Smokers report that they often smoke cigarettes during stressful times. Smoking and stress produce similar physiological responses such as increases in heart rate, blood pressure, and adrenaline levels. The combination of smoking and stress results in greater increases in these physiological responses compared to smoking or stress alone. Such increases are thought to be harmful to cardiovascular health. Additionally, smokers with exaggerated responses to stress may be more likely to relapse following a smoking cessation attempt. The purpose of this study is to assess the effects of paroxetine, a selective serotonin reuptake inhibitor (SSRI), on the cardiovascular response to stress after smoking.

Participants in this double-blind, placebo-controlled study will receive 1 month of paroxetine and 1 month of placebo with the order of which is taken during the first month randomly assigned. Paroxetine will be administered at a daily dose of 10 mg for the first week and increased to a daily dose of 20 mg for the remainder of the study. After one month of medication, participants will abstain from smoking for one night and then undergo mental stress testing the following day. Immediately prior to the mental stress testing, participants will smoke a cigarette. Mental stressors will include speaking and math tasks. Physiological measures of stress (e.g., blood pressure, heart rate, and plasma catecholamine concentrations) and subjective measures of stress will be evaluated. Following the second month of medication, participants will again undergo the procedure for mental stress testing and evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Smokes an average of at least 10 cigarettes per day during the year prior to enrollment

Exclusion Criteria:

* Interested in quitting smoking within the 3 months following enrollment
* Current unstable medical condition
* Substance abuse within the year prior to enrollment
* Current use of any medications (e.g., psychoactive medications, antihypertensives) that, in the opinion of the investigators, might interfere with study measures or that would be expected to interact with paroxetine (e.g., CYP2D6 substrates)
* Smoking cessation therapy within the 3 months prior to enrollment
* Regular use of any form of tobacco other than cigarettes
* Significant psychiatric disorders as assessed by the PRIME-MD and verified by a clinician
* History of hypersensitivity to any selective serotonin reuptake inhibitor
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2005-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kotlyar, Principal Investigator — University of Minnesota
Locations (1):
- College of Pharmacy, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Kotlyar M, al'Absi M, Thuras P, Vuchetich JP, Adson DE, Nowack AL, Hatsukami DK. Effect of paroxetine on physiological response to stress and smoking. Psychosom Med. 2013 Apr;75(3):236-43. doi: 10.1097/PSY.0b013e3182898f6d. Epub 2013 Mar 15. PMID 23504241

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (4 Weeks) Then Paroxetine (4 Weeks): Placebo once daily in first intervention period and Paroxetine 10 mg daily for 1 week then increased to 20 mg once daily for remainder of second intervention period
- Paroxetine (4 Weeks) the Placebo (4 Weeks): Paroxetine 10 mg daily for 1 week then increased to 20 mg once daily for remainder of first intervention period, placebo once daily in second intervention period
Period: First Intervention (4 Weeks)
Arm/Group | Placebo (4 Weeks) Then Paroxetine (4 Weeks) | Paroxetine (4 Weeks) the Placebo (4 Weeks)
Started | 58 | 47
Completed | 40 | 35
Not Completed | 18 | 12
Period: Second Intervention (4 Weeks)
Arm/Group | Placebo (4 Weeks) Then Paroxetine (4 Weeks) | Paroxetine (4 Weeks) the Placebo (4 Weeks)
Started | 40 | 35
Completed | 33 | 30
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Population: Includes subjects who completed both laboratory sessions (n=62). One additional subject completed both laboratory sessions but did not have usable measures in the primary outcomes (cardiovascular measures) and was excluded
Groups:
- Placebo First 4 Weeks, Then Paroxetine for 4 Weeks: Placebo once daily in first intervention period and Paroxetine 10 mg daily for 1 week then increased to 20 mg once daily for remainder of second intervention period
- Paroxetine First 4 Weeks, Then Placebo for 4 Weeks: Paroxetine 10 mg daily for 1 week then increased to 20 mg once daily for remainder of first intervention period, placebo once daily in second intervention period
- Total: Total of all reporting groups
Arm/Group | Placebo First 4 Weeks, Then Paroxetine for 4 Weeks | Paroxetine First 4 Weeks, Then Placebo for 4 Weeks | Total
Number analyzed (Participants) | 33 | 29 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 29 | 62
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (14.1) | 40.0 (11.0) | 40.2 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 17 | 15 | 32
Region of Enrollment [Number; unit: participants]
  United States | 33 | 29 | 62

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure Response to Stress
Description: Change in systolic blood pressure from Resting period to that observed during a speech delivered immediately after smoking a cigarette
Time Frame: After 4 weeks of paroxetine / placebo
Measure: Mean (Standard Error); unit: mmHg
Groups:
- After 4 Weeks of Placebo: Change in systolic blood pressure from Resting period to that observed during a speech delivered immediately after smoking a cigarette in those receiving 4 weeks of placebo
- After 4 Weeks of Paroxetine: Change in systolic blood pressure from Resting period to that observed during a speech delivered immediately after smoking a cigarette in those receiving 4 weeks of paroxetine (1 week of 10 mg once daily followed by 3 weeks of 20 mg once daily)
Arm/Group | After 4 Weeks of Placebo | After 4 Weeks of Paroxetine
Number analyzed (Participants) | 62 | 62
mmHg | 16.85 (0.78) | 11.71 (0.78)
Statistical Analysis 1: Comparison: After 4 Weeks of Placebo vs After 4 Weeks of Paroxetine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

2. Other Pre Specified Outcome: Diastolic Blood Pressure Response to Stress
Description: Change in diastolic blood pressure from Resting period to that observed during a speech delivered immediately after smoking a cigarette
Time Frame: After 4 weeks of paroxetine / placebo
Measure: Mean (Standard Error); unit: mm Hg
Groups:
- After 4 Weeks of Placebo: Change in diastolic blood pressure fom Resting period to that observed during a speech delivered immediately after smoking a cigarette in those receiving 4 weeks of placebo
- After 4 Weeks of Paroxetine: Change in diastolic blood pressure from Resting period to that observed during a speech delivered immediately after smoking a cigarette in those receiving 4 weeks of paroxetine (1 week of 10 mg once daily followed by 3 weeks of 20 mg once daily)
Arm/Group | After 4 Weeks of Placebo | After 4 Weeks of Paroxetine
Number analyzed (Participants) | 62 | 62
mm Hg | 9.78 (0.49) | 8.07 (0.5)
Statistical Analysis 1: Comparison: After 4 Weeks of Placebo vs After 4 Weeks of Paroxetine; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis

3. Other Pre Specified Outcome: Heart Rate Response to Stress
Description: Change in heart rate from Resting period to that observed during a speech delivered immediately after smoking a cigarette
Time Frame: After 4 weeks of paroxetine / placebo
Measure: Mean (Standard Error); unit: beats/minute
Groups:
- After 4 Weeks of Placebo: Change in heart rate from Resting period to that observed during a speech delivered immediately after smoking a cigarette in those receiving 4 weeks of placebo
- After 4 Weeks of Paroxetine: Change in heart rate from Resting period to that observed during a speech delivered immediately after smoking a cigarette in those receiving 4 weeks of paroxetine (1 week of 10 mg once daily followed by 3 weeks of 20 mg once daily)
Arm/Group | After 4 Weeks of Placebo | After 4 Weeks of Paroxetine
Number analyzed (Participants) | 62 | 62
beats/minute | 20.39 (0.56) | 20.02 (0.56)
Statistical Analysis 1: Comparison: After 4 Weeks of Placebo vs After 4 Weeks of Paroxetine; Test type: Superiority or Other; p = 0.56, Mixed Models Analysis

4. Other Pre Specified Outcome: Plasma Epinephrine Concentration Response to Stress
Description: Change in plasma epinephrine concentrations from Resting period to those observed during a speech delivered immediately after smoking a cigarette
Time Frame: After 4 weeks of paroxetine / placebo
Measure: Mean (Standard Error); unit: pg / ml
Groups:
- After 4 Weeks of Placebo: Change in plasma epinephrine concentrations from Resting period to those observed during a speech delivered immediately after smoking a cigarette in those receiving 4 weeks of placebo
- After 4 Weeks of Paroxetine: Change in plasma epinephrine concentrations from Resting period to those observed during a speech delivered immediately after smoking a cigarette in those receiving 4 weeks of paroxetine (1 week of 10 mg once daily followed by 3 weeks of 20 mg once daily)
Arm/Group | After 4 Weeks of Placebo | After 4 Weeks of Paroxetine
Number analyzed (Participants) | 62 | 62
pg / ml | 40.98 (3.42) | 34.94 (3.48)
Statistical Analysis 1: Comparison: After 4 Weeks of Placebo vs After 4 Weeks of Paroxetine; Test type: Superiority or Other; p = 0.33, Mixed Models Analysis

5. Other Pre Specified Outcome: Plasma Norepinephrine Concentration Response to Stress
Description: Change in plasma norepinephrine concentrations from Resting period to those observed during a speech delivered immediately after smoking a cigarette
Time Frame: After 4 weeks of paroxetine / placebo
Measure: Mean (Standard Error); unit: pg / ml
Groups:
- After 4 Weeks of Placebo: Change in plasma norepinephrine concentrations from Resting period to those observed during a speech delivered immediately after smoking a cigarette in those receiving 4 weeks of placebo
- After 4 Weeks of Paroxetine: Change in plasma norepinephrine concentrations from Resting period to those observed during a speech delivered immediately after smoking a cigarette in those receiving 4 weeks of paroxetine (1 week of 10 mg once daily followed by 3 weeks of 20 mg once daily)
Arm/Group | After 4 Weeks of Placebo | After 4 Weeks of Paroxetine
Number analyzed (Participants) | 62 | 62
pg / ml | 72.31 (18.32) | 63.37 (18.32)
Statistical Analysis 1: Comparison: After 4 Weeks of Placebo vs After 4 Weeks of Paroxetine; Test type: Superiority or Other; p = 0.82, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse events data collected during treatment (i.e. 4 weeks of paroxetine or 4 weeks of placebo)
Description: Subjects were asked at each visit an open ended question if they've experienced any side effects
Groups:
- During 4 Weeks of Placebo: Participants receive placebo daily for 4 weeks
- During 4 Weeks of Paroxetine: Participants received paroxetine 10 mg once daily for 1 week followed by 20 mg once daily for 3 weeks
Arm/Group | During 4 Weeks of Placebo | During 4 Weeks of Paroxetine
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 34/62 | 35/62
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | During 4 Weeks of Placebo (N=62) | During 4 Weeks of Paroxetine (N=62)
Dizziness (General disorders) | 1 | 6
Gastrointenstinal symptoms (Gastrointestinal disorders) | 7 | 13
drowsiness (General disorders) | 10 | 16
sexual side effects (Reproductive system and breast disorders) | 1 | 5
insomnia (General disorders) | 3 | 4
dry mouth / taste changes (General disorders) | 1 | 6
headache (General disorders) | 1 | 4
change in appetite (Gastrointestinal disorders) | 5 | 3
unusual dreams (General disorders) | 5 | 0
anxiety / irritability (General disorders) | 8 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No